CLINICAL TRIAL: NCT03962218
Title: Randomized Controlled Trial to Assess the Effectiveness of Aquatic Specific Physiotherapy in the Improvement of Balance and Gait.
Brief Title: Aquatic Specific Physiotherapy on Incomplete Spinal Cord Injuries
Acronym: FALMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ECA-FALMI-19
Record Dates: First submitted 2019-05-14; First posted 2019-05-23 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Spinal Cord Injuries
Keywords: spinal cord injury; Hydrotherapy; Balance; Gait
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Hydrotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Aquatic Therapy (EAT) (Experimental): Aquatic physiotherapy treatment at time 1 (week 1)
  Interventions: Procedure: aquatic physiotherapy
- Late Aquatic Therapy (LAT) (Other): Control for Group 1 for the 5 first weeks of Group 1 treatment. Aquatic physiotherapy treatment at time 2 (week 6).
  Interventions: Procedure: aquatic physiotherapy

INTERVENTIONS:
Procedure: aquatic physiotherapy — specific aquatic physiotherapy 3 times a week, for 6 weeks, including feet balance exercises (Rating of Perceived Effort (RPE)), slow walking in all directions, walking with obstacles, Ai Chi, exercises of muscular strength. Each session duration is of 40 minutes.
  Other Names: hydrotherapy

SUMMARY:
Purpose of the study: To analyse the effectiveness of aquatic physiotherapy on spinal cord injuries (LMi) in the improvement of balance and gait, in the inflammatory profile, and the impact on the quality of life.

Main objective: To analyse if there are differences in the recovery of the balance, in incomplete subacute spinal cord injuries, with lesion level T1-L5 and ASIA (American Spinal Injury Association) C and D .

Secondary objectives:

1. functional gait
2. To evaluate if the time from the injury to the start of the aquatic therapy influences the results on balance and functional gait.
3. To study the effect of aquatic therapy on serum markers of systemic inflammation.
4. Quality of life related to health. Design: Crossed, controlled and randomized clinical trial, with blind evaluation of the response variables.

Scope of the study: National Hospital of Paraplegics. Toledo (Spain). Population: Subjects with incomplete spinal cord injury ASIA C and D. n = 50 (25 in each arm randomly).

Intervention:

6 weeks of specific Aquatic Physiotherapy (3 times a week). Group 1 will perform aquatic physiotherapy at the time of entering the study, and group 2 will perform it 6 weeks later.

Outcomes: Static and dynamic balance (Berg test and Time Up and Go). Speed of the gait (test of 10 m.). Gait resistance (6 min. Test). Functional capacity of the gait (WISCI II). Biomechanical analysis (sensorial-dynamic, rhythmic and directional control, and gait test) by posturography. Questionnaires EuroQol-5Dimensions-5Level (EQ-5D-5L) and the Spanish Version of the Quality of Life Index (SV-QLI) in spinal cord injury (SCI).

Biomarkers of inflammation: 20 cytokines. Analysis of results: The main outcome measure will be the percentage of patients who have improved. Considering improvement when the difference between the groups is, at least, a 10% of their score in the Berg test between V0 and V1 (with their corresponding 95% confidence intervals). It will be adjusted for confounding and interaction factors with a multivariate analysis using logistic regression. All analyses will be performed according to the intention to treat principle.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with incomplete spinal cord injury T1-L5 (ASIA C y D).
* Traumatic and not traumatic injuries, with injury date of less than 8 months.
* Able to maintain assisted standing up
* Subjects signing the informed consent form

Exclusion Criteria:

* Subjects with progressive injuries.
* heart or lung disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
balance | 12 weeks
  Berg test
Speed of the gait | 12 weeks
  test of 10 m
Gait resistance | 12 weeks
  6 Minutes Walk Test
Functional capacity of the gait | 12 weeks
  Walking Index for spinal cord injury (WISCI II)

SECONDARY OUTCOMES:
General quality of life related to Health | 12 weeks
  Measures through the Questionnaire EuroQol-5D-5L. The questionnaire comprises 5 dimensions: mobility, self care, usual activities, pain discomfort, anxiety/depression. Each dimension is scored in 5 levels, 1-5 (level 1-no problem, level 5,-extreme problems). Based on the answers, a index value from 0 to 1 is calculated (0-the worst quality of life, 1-the best quality of life).
Specific quality of life related to health in spinal cord injury | 12 weeks
  Measured through the questionnaire "Spanish version of the Quality of Life Index in spinal cord injury (SV-QLI / SCI)". The questionnaire evaluates 37 items, in a scale from 1 (less satisfied) to 6 (most satisfied). There are 5 scores of 0-30 (0=less satisfied, 30=most satisfied) which are calculated using the subscales: 1-Total Quality of Life score. 2-Health and Functioning Subscale. 3-Social and Economic Subscale. 4-Psychological /Spiritual Subscale. 5-Family Subscale. The final score is an average of the subscale's scores, being between 0 (0=less satisfied) and 30 (30=most satisfied).
Inflammatory cytokines analysis | 12 weeks
  Quantification of the cytokine concentration, in pg/mL, will be carried out by Luminex xMAP Bead-based multiplex Assay (Labclinics). Cytokine's panel includes the cytokines E-selectin, P-selectin, IL-1α, IL-1β, IL-10, MCP-1 (CCL2),GM-CSF, IL12p70, MIP-1α (CCL3), MIP-1β (CCL4), ICAM-1, IL-4, IL-13, IFN-α, IFN-γ, IL-6, IL-17A,(CTLA8), IL-8 (CXCL8), IP-10 (CXCL10) and TNF-α.

CONTACTS AND LOCATIONS:
Overall Officials: Inés Martínez-Galán, MD, Principal Investigator — University of Castilla-La Mancha
Locations (1):
- Hospital Nacional de Parapléjicos, Toledo, Spain

REFERENCES:
- [Derived] Menchero R, Martinez-Galan I, Alcobendas-Maestro M, Romay-Barrero H, Fernandez-Maestra A, Gueita-Rodriguez J. Feasibility and impact of a Water Specific Therapy program in individuals with subacute incomplete spinal cord injury: A non-randomized controlled trial. J Spinal Cord Med. 2025 Nov;48(6):997-1005. doi: 10.1080/10790268.2025.2472098. Epub 2025 Mar 31. PMID 40163138